CLINICAL TRIAL: NCT01549626
Title: Effects of Flaxseed Flour - Whole Brown Flaxseed Flour, Brown Defatted Flaxseed Flour and Golden Flaxseed Flour in Appetite Sensations Satiety, Lipid Profile, Pressure Levels and Associated Costs Among Overweighed and Obese Women
Brief Title: Effects of Flaxseed Flour in Appetite Sensations, Lipid Profile and Pressure Levels Among Overweighed and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Wania Lucia Araujo Monteiro, Nutritionist, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: w831102m
Record Dates: First submitted 2012-02-28; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Adult Women; Overweight; Obese
Keywords: Flaxseed; Women; Obesity; No smokers
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- defatted flaxseed flour (Active Comparator): 30 grams per day of defatted flaxseed flour
  Interventions: Dietary Supplement: Golden flaxseed flour; Dietary Supplement: Whole brown flaxseed flour
- golden flaxseed flour (Active Comparator): 30 grams per day of golden flaxseed flour
  Interventions: Dietary Supplement: Defatted flaxseed flour; Dietary Supplement: Whole brown flaxseed flour
- whole brown flaxseed flour (Active Comparator): 30 grams per day of whole brown flaxseed flour
  Interventions: Dietary Supplement: Defatted flaxseed flour; Dietary Supplement: Golden flaxseed flour

INTERVENTIONS:
Dietary Supplement: Defatted flaxseed flour — 30g defatted flaxseed flour per day for breakfast
  Other Names: Golden flaxseed flour; Whole brown flaxseed flour
  Arms: golden flaxseed flour; whole brown flaxseed flour
Dietary Supplement: Golden flaxseed flour — 30 grams of golden flaxseed flour per day for breakfast
  Other Names: Defatted flaxseed flour; Whole brown flaxseed flour
  Arms: defatted flaxseed flour; whole brown flaxseed flour
Dietary Supplement: Whole brown flaxseed flour — 30 grams of whole brown flaxseed flour per day for breakfast
  Other Names: Defatted flaxseed flour; Golden flaxseed flour
  Arms: defatted flaxseed flour; golden flaxseed flour

SUMMARY:
Inclusion of foods rich in fiber, such as flaxseed, is a nutritional strategy for treating obesity. The hypothesis of this study is to compare the effects of three types of flaxseed flour - whole brown flaxseed flour, brown defatted flaxseed flour and golden flaxseed flour in the sensations of appetite and satiety, lipid profile, pressure levels and associated costs in overweight and obese women.

ELIGIBILITY:
Inclusion Criteria:

* adult women

Exclusion Criteria:

* women diabetic
* menopausal
* smokers
* pregnant
* using anorectic and satiogenic drugs

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Appetite | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF), and golden flaxseed flour (GFF) - in subjective sensations of appetite in overweighed and obese women.

SECONDARY OUTCOMES:
Satiety | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF), and golden flaxseed flour (GFF) - in subjective sensations of satiety in overweighed and obese women.
LDL-cholesterol | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF) and golden flaxseed flour (GFF) - in reducing cardiovascular risk factors in overweighed and obese women.
HDL-cholesterol | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF) and golden flaxseed flour (GFF) - in reducing cardiovascular risk factors in overweighed and obese women.
Total Cholesterol | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF) and golden flaxseed flour (GFF) - in reducing cardiovascular risk factors in overweighed and obese women.
Triglycerides | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF) and golden flaxseed flour (GFF) - in reducing cardiovascular risk factors in overweighed and obese women.
Glucose | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF) and golden flaxseed flour (GFF) - in reducing cardiovascular risk factors in overweighed and obese women.
Uric acid | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF) and golden flaxseed flour (GFF) - in reducing cardiovascular risk factors in overweighed and obese women.
Systemic blood pressure | Up to 2 months
  Compare the effects of three different types of flaxseed flour - whole brown flaxseed flour (WBFF), brown defatted flaxseed flour (BDFF) and golden flaxseed flour (GFF) - in reducing cardiovascular risk factors in overweighed and obese women.

CONTACTS AND LOCATIONS:
Locations (1):
- Clementino Fraga Filho University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil